CLINICAL TRIAL: NCT04256902
Title: Self-identification Based Intervention Targeting Sexual Orientation and Gender Identity
Brief Title: Lesbian, Gay, Bisexual, and Transgender (LGBT) Conference
Acronym: LGBT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0069
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Lesbian; Gay; Bisexual; Transgender
Keywords: self-identification; discrimination; mental health
MeSH Terms: conditions — Homosexuality, Female; Homosexuality; Bisexuality; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite increased visibility and acceptance of the LGBT community (Lesbian, Gay, Bisexual and Transgender), in some parts of society, many LGBT people struggle with self-acceptance. Minority Stress Theory, described in the scientific literature, explains that health disparities among populations such as the LGBT population can be explained by stressors induced by a hostile, homophobic culture, which results in harm suffered, expectations of rejection, and internalized homophobia. The harm suffered may include acts of discrimination, harassment, violence (physical or linguistic). But more deeply, two important points of this theory: 1) the expectations of the LGBT person to experience rejection based on their identity and the anti-LGBT social stigma, 2) internalized homophobia, which is a social internalization from negativity against homosexuality and transgender to the initial stages of the identity development of an individual who can continue throughout his life. Perceived harm, stigma and lived rejection are associated with an increased propensity to experience significant psychological pain. LGBT people are more likely to develop self-identification based on sexual orientation or gender, making them more vulnerable to any rejection signal.

There is a growing scientific interest around Cognitive and Behavioral Therapies (CBT) of 3rd wave, also called therapies derived from Buddhism, or therapies based on meditation. These programs aim to observe and test, through an experiential meta-cognitive practice, the dogmas or preconceptions (about ourselves, others, and the world) and mental attitudes that guide our choices without our knowledge and are at the origin of suffering, in order to gain inner freedom. These practices constitute an experiential scientific methodology of self-knowledge and reality. These secular programs have become a standard treatment in the management of stress, chronic pain, and the prevention of relapsing depression. In addition, the interest of these practices has been demonstrated in many areas of somatic and psychiatric medicine (including depression and suicidal behavior), but also for the promotion of mental health in the general population. This topic is the subject of more than 15,000 international scientific publications with reading committee (Medline indexed), and of strong interest and shared by both the scientific community and the general public.

Scientists are currently deepening these therapies with a focus on wisdom-based self-identification. Beyond the name "therapies", this educational information is key to life for everyone. Who am I ? Am I defined by my social roles, my physical characteristics, my preferences? How to face external challenges? How to develop real self-confidence?

Dr Déborah Ducasse offers a conference on the theme: "Sexual orientation, gender: where is the problem?" Nowhere. Self-identification. ". This conference will take place on 05/15/2020, on the occasion of World Day Against Homophobia.

In line with the OECD press release in 2019 "The LGBT challenge: how to improve the integration of sexual and gender minorities? "(Panorama de la société 2019: Social Indicators of the OECD), the investigators want to assess whether an intervention targeting valid self-identification can 1) have a positive impact on the acceptance and discrimination indicators of the OECD ; 2) have an impact on valid self-identification.

Direct benefits are expected, psychologically and socially, in the fight against discrimination, inclusion and self-acceptance.

In the medium and long term: major public health interest via the adaptation of psychoeducational interventions based on self-identification in order to prevent psychosocial risks and suicidal behavior in connection with an altered self-identification based on sexual orientation and gender.

DETAILED DESCRIPTION:
A wide communication (media, social networks) will be organized around this conference which is free to enter A prior registration will be requested by email. For each person sending an email to register, they will be offered to participate in the research by following the web link to the Google Form questionnaire ("pre-conference") with information on the proposed research. Refusal to participate in the research will not prevent you from attending the conference, this will be mentioned when sending the link to the questionnaire.

At the end of the conference, another email will be sent to those who have agreed to participate with a new Google Form link to answer specific "post-conference" questions.

The impact of the conference will be studied by comparing the pre and post conference questionnaires

Main objective: Evaluate the impact of an educational intervention on self-identification (conference "Sexual orientation, gender: where is the problem? Nowhere. Self-identification." Lasting 2 hours), on the acceptance of homosexuality and transgender, in people coming to attend this intervention (evaluations before and after)

Secondary objectives: Evaluate the impact of an educational intervention on self-identification (2 hours), on the representations of stigmatization of homosexuality and transgender, in people coming to attend this intervention (evaluations before- after).

ELIGIBILITY:
Inclusion criteria:

- be registered for the LGBT conference

Exclusion criteria

* Subject unable to read or/and write

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all those registered for the conference and who agree to participate by answering the questionnaires
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
acceptance of LGBT | 1 day
  Criteria for assessing acceptance as mentioned in the 2019 OECD report

SECONDARY OUTCOMES:
stigmatisation of LGBT | 1 day
  Criteria for assessing acceptance as mentioned in the 2019 OECD report

CONTACTS AND LOCATIONS:
Overall Officials: DEBORAH DUCASSE, MD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC